CLINICAL TRIAL: NCT04757220
Title: Cognitive and Neural Mechanisms of Multidimensional Apathy in Psychiatric Pathologies
Brief Title: Multidimensional Apathy in Psychiatric Pathologies.
Acronym: AmSeD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 8062
Record Dates: First submitted 2021-01-12; First posted 2021-02-17 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Apathy
MeSH Terms: conditions — Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with schizophrenia (Experimental): * 5 subjective questionnaires
  * 4 cognitive tasks with EEG recordings
  Interventions: Other: Cognitive tasks with EEG recording
- Patients with depression (Experimental): * 5 subjective questionnaires
  * 4 cognitive tasks with EEG recordings
  Interventions: Other: Cognitive tasks with EEG recording
- Healthy controls (Active Comparator): * 5 subjective questionnaires
  * 4 cognitive tasks with EEG recordings
  Interventions: Other: Cognitive tasks with EEG recording

INTERVENTIONS:
Other: Cognitive tasks with EEG recording — questionnaires and cognitives tasks

SUMMARY:
Apathy is defined by quantitative decrease in goal-directed activity in comparison to the person's previous level of functioning. Apathy is a transnosographic symptom, prevalent in many neurological and psychiatric pathologies (specifically in schizophrenia and depression), and almost half of patients suffer from it. It is an important source of burden, affecting both personal and occupational life. Despite its high prevalence and negative consequences, no pharmacological or non-pharmacological treatments exist, the underlying mechanisms of apathy being poorly understood. The main aim of the present study is to advance in our knowledge of cognitive and neural mechanisms of apathy by using a multidimensional model of apathy, distinguishing three forms: executive, emotional and auto-activation/initiative.

the investigators hypothesize, independently of the pathology (schizophrenia and depression), the existence of different cognitive deficits underlying each of the 3 subforms of apathy. Indeed, according to the predictions of Levy and Dubois' model (2006), executive disorders underlie the cognitive form of apathy. It may be related to lesions of the dorsolateral prefrontal cortex and the cognitive territory of the basal ganglia. Emotional apathy could be due to motivational disorder. Dysfunctions or lesions in the orbital and medial prefrontal cortex and limbic territories of the basal ganglia may underlie this. Finally, the initiative form, may be a mixed form, with both motivational and executive difficulties. Lesions or dysfunctions may affect both the cognitive and limbic territories of the basal ganglia or the anterior cingulate cortex.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria (all subjects):
* age between 18 and 60 years
* men or women volunteers, hospitalized or not
* subject affiliated to an health insurance
* subject having signed an informed consent

Inclusion criteria (for schizophrenic patients):

- presence of DSM-V TR criteria for schizophrenia (American Psychiatric Association, 1994)

Inclusion criteria (for depressive patients):

- presence of DSM-V TR criteria for depression (American Psychiatric Association, 1994)

Exclusion Criteria:

* a major or non stabilized somatic disorder
* medical history likely to affect cerebral anatomy or linked to an abnormality (neonatal distress, neurochirurgical intervention, neurological disorders, stroke attack)
* any disorders involved in the use of a psycho-active substance (as defined by the DSM-IV)
* sensory disabling impairments, and specifically visual acuity < 8
* general anaesthesia during the 3 months before the study
* pregnancy (declared by the subject)
* persons in an emergency situation
* persons deprived in any way of their liberty
* persons in period of exclusion in an other protocol

Exclusion criteria (for controls):

- use of psychotropic substance during the 3 weeks before the study

Exclusion criteria (for patients):

- use of benzodiazepines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the motivational form of apathy | first baseline visit
  The severity of the forms of apathy (Executive, Emotive and Initiation apathy) will be measured by using The Dimensional Apathy Scale (DAS) (Radakovic and Abrahams, 2014) and the Lille Apathy Rating Scale (LARS) (Sockeel et al., 2006) Items are scored on a 4-point Likert scale based on the frequency of occurrence of the apathetic symptoms in the previous month. 3 scores will be obtained, one for each form of apathy. A high score (maximum, 24) indicates a severe form of apathy.
Assessment of the cognitive form of apathy | first baseline visit
  The severity of the forms of apathy (Executive, Emotive and Initiation apathy) will be measured by using The Dimensional Apathy Scale (DAS) (Radakovic and Abrahams, 2014) and the Lille Apathy Rating Scale (LARS) (Sockeel et al., 2006) Items are scored on a 4-point Likert scale based on the frequency of occurrence of the apathetic symptoms in the previous month. 3 scores will be obtained, one for each form of apathy. A high score (maximum, 24) indicates a severe form of apathy.
Assessment of the behavioural form of apathy | first baseline visit
  The severity of the forms of apathy (Executive, Emotive and Initiation apathy) will be measured by using The Dimensional Apathy Scale (DAS) (Radakovic and Abrahams, 2014) and the Lille Apathy Rating Scale (LARS) (Sockeel et al., 2006) Items are scored on a 4-point Likert scale based on the frequency of occurrence of the apathetic symptoms in the previous month. 3 scores will be obtained, one for each form of apathy. A high score (maximum, 24) indicates a severe form of apathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No